CLINICAL TRIAL: NCT03750643
Title: Phase 1, Multicenter, Randomized, Placebo-Controlled, Triple-Blind, Single-Ascending Dose and Repeat-Dose Trial in Healthy Participants and Participants With Atopic Dermatitis
Brief Title: A Study of LY3454738 in Healthy Participants and Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17090; J1B-MC-FRCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3454738 - Part A (Experimental): Escalating doses of LY3454738 administered intravenously (IV) or subcutaneously (SC) to healthy participants
  Interventions: Drug: LY3454738
- Placebo - Part A (Placebo Comparator): Placebo administered IV to healthy participants
  Interventions: Drug: Placebo
- LY3454738 - Part B (Experimental): LY3454738 administered IV to healthy participants
  Interventions: Drug: LY3454738
- Placebo - Part B (Placebo Comparator): Placebo administered IV to healthy participants
  Interventions: Drug: Placebo
- LY3454738 - Part C (Experimental): LY3454738 administered IV to participants with atopic dermatitis (AD)
  Interventions: Drug: LY3454738
- Placebo - Part C (Placebo Comparator): Placebo administered IV to participants with AD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3454738 — Administered IV
  Arms: LY3454738 - Part A; LY3454738 - Part B; LY3454738 - Part C
Drug: LY3454738 — Administered SC
  Arms: LY3454738 - Part A
Drug: Placebo — Administered IV
  Arms: Placebo - Part A; Placebo - Part B; Placebo - Part C

SUMMARY:
The main purpose of this study is to investigate the safety, tolerability, and efficacy of the study drug known as LY3454738 in healthy participants and participants with atopic dermatitis. The study has three parts. Each participant will enroll in one part. The study will last 12 to 24 weeks, depending on part.

ELIGIBILITY:
Inclusion Criteria:

* All: Must have a body mass index of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive, for Parts A and B, and 18.0 to 45.0 kg/m², inclusive, for Part C and a minimum body weight of 50 kilograms
* For PART A and B only, regarding the inclusion of healthy Japanese participants: Minimum age is 20 years and the participant's biological parents and all of the participant's biological grandparents must be of exclusive Japanese descent and must have been born in Japan
* AD:

  * Must have a diagnosis of AD for at least 12 months with either poor response to topical treatments or inability to use topical treatments
  * Must agree to use moisturizer daily throughout the treatment period

Exclusion Criteria:

* All: must not have previously completed a clinical trial with a molecule targeting interleukin-33 (IL-33) or its receptor
* AD:

  * Must not have received certain topical medications for AD within 2 weeks prior to randomization
  * Must not have received certain oral medications for AD or received phototherapy within 4 weeks prior to randomization
  * Must not have received any antibody-based biologic agents (marketed or investigational) within 5 half lives (t1/2) of the drug prior to randomization
  * Must not have received intravenous, intramuscular, or intra-articular steroids in the past 6 weeks prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 24
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Number of Participants Achieving a Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) Score of 0 or 1 with a ≥ 2-point Improvement from Baseline | Week 12
  The vIGA-AD measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) of LY3454738 | Day 1 through Day 85 (Day 99 for Part C)
  Cmax of LY3454738
Area Under the Concentration-Versus-Time Curve (AUC) of LY3454738 | Day 1 through Day 85 (Day 99 for Part C)
  AUC of LY3454738

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (19):
  - Pinnacle Research Group, Anniston, Alabama
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - California Clinical Trials Medical Group, Glendale, California
  - Revival Research Corporation, Doral, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Skin Sciences, PLLC, Louisville, Kentucky
  - PAREXEL-Phase 1 Baltimore Harbor Hospital Center, Baltimore, Maryland
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - JUVA Skin & Laser Center, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Wright State Physicians Dermatology, Dayton, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Premier Clinical Research, Spokane, Washington
- Puerto Rico (2):
  - Dermatology, Los Prados, Caguas
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3454738 in Healthy Participants and Participants With Atopic Dermatitis (Eczema) — https://trials.lillytrialguide.com/en-US/trial/1FiRtIYceUkw4QOKAMusai